CLINICAL TRIAL: NCT02308826
Title: Multi-Component Early Intervention for Socially Inhibited Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Andrea Chronis-Tuscano, Professor, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH103253-01A1 (NIH)
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Behavioral Inhibition; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Turtle Program (Experimental): The Turtle Program involves a child social and emotional skills group (Social Skills Facilitated Play) and a modification of Parent-Child Interaction Therapy in which parents are provided in-vivo coaching in following their children's lead and encouraging approach behaviors within the peer context. The child group provides a forum of same-age peers to learn to develop social and emotion regulation skills. The Turtle Program is administered over an 8-week period.
  Interventions: Behavioral: Turtle Program
- Cool Little Kids (Active Comparator): A 6-week parent psychoeducation group administered over an 8-week period.
  Interventions: Behavioral: Cool Little Kids

INTERVENTIONS:
Behavioral: Turtle Program
  Arms: Turtle Program
Behavioral: Cool Little Kids
  Arms: Cool Little Kids

SUMMARY:
This project is intended to provide a rigorous test of the Turtle Program, an early intervention program for behaviorally inhibited preschoolers. The proposed project will extend promising pilot study findings by: (a) evaluating the integrated intervention in a larger sample (n = 150) of 45-64 month children and their parents, which will allow for an examination of mediators and moderators of treatment effects; (b) comparing the Turtle Program to the best available treatment for preschool behavioral inhibition, the Cool Little Kids (CLK) parent psychoeducation group; (c) examining heart rate reactivity and regulation as both baseline moderators of treatment response and as outcome measures; (d) examining parent anxiety disorders as a moderator of treatment response; (e) including a mid-treatment assessment and extending follow-up to one year.

ELIGIBILITY:
Inclusion Criteria:

* child must be attending preschool; child must score within top 15% on parent-rated Behavioral Inhibition Questionnaire

Exclusion Criteria:

* child has a diagnosis of pervasive developmental disorder, selective mutism, or mental retardation; child scores above clinical cutoff on Social Communication Questionnaire; child is currently receiving treatment for anxiety; child does not have a custodial parent who has also consented to participate

Ages: 45 Months to 64 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 169 (Actual)
Dates: Start 2014-12; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in child anxiety disorder symptoms | pre-treatment, mid-treatment (week 4), post-treatment (week 8), and 1-year follow-up
  Assessed with diagnostic interviews (Anxiety Disorders Interview Schedule) with parents

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Chronis-Tuscano, Ph.D., Principal Investigator — University of Maryland; Kenneth Rubin, Ph.D., Principal Investigator — University of Maryland
Locations (1):
- Maryland ADHD Program, College Park, Maryland, United States

REFERENCES:
- [Derived] Fleece H, Wagner NJ, Chronis-Tuscano A, Smith KA, Novick DR, Druskin LR, Shakiba N, Danko CM, Rubin KH. Can behaviorally inhibited preschoolers make friends? Dev Psychol. 2024 Jul;60(7):1203-1213. doi: 10.1037/dev0001742. Epub 2024 Apr 22. PMID 38647467
- [Derived] Novick DR, Meyer CT, Wagner NJ, Rubin KH, Danko CM, Dougherty LR, Druskin LR, Smith KA, Chronis-Tuscano A. Testing reciprocal associations between child anxiety and parenting across early interventions for inhibited preschoolers. J Child Psychol Psychiatry. 2023 Dec;64(12):1665-1678. doi: 10.1111/jcpp.13879. Epub 2023 Aug 29. PMID 37644651
- [Derived] Wagner NJ, Shakiba N, Bui HNT, Sem K, Novick DR, Danko CM, Dougherty LR, Chronis-Tuscano A, Rubin KH. Examining the Relations Between Children's Vagal Flexibility Across Social Stressor Tasks and Parent- and Clinician-Rated Anxiety Using Baseline Data from an Early Intervention for Inhibited Preschoolers. Res Child Adolesc Psychopathol. 2023 Aug;51(8):1213-1224. doi: 10.1007/s10802-023-01050-3. Epub 2023 Mar 24. PMID 36961596
- [Derived] Chronis-Tuscano A, Novick DR, Danko CM, Smith KA, Wagner NJ, Wang CH, Druskin L, Dougherty LR, Rubin KH. Early intervention for inhibited young children: a randomized controlled trial comparing the Turtle Program and Cool Little Kids. J Child Psychol Psychiatry. 2022 Mar;63(3):273-281. doi: 10.1111/jcpp.13475. Epub 2021 Jun 29. PMID 34184792